CLINICAL TRIAL: NCT05251506
Title: The Evaluation of Laser Lancing Devices in Constructing Self-management Systems for Chronic Diseases in Adult Diabetes Patients
Brief Title: The Evaluation of Laser Lancing Devices in Adult Type 2 Diabetes Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Korea University Guro Hospital (Other)
Collaborators: Korea Medical Device Development Fund (Unknown)
Responsible Party: Principal Investigator, Hye Jin Yoo, Professor, Korea University Guro Hospital
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: K2021-1520-002
Record Dates: First submitted 2021-09-02; First posted 2022-02-22 (Actual); Last update posted 2022-02-22 (Actual); Status verified 2022-02

CONDITIONS: Type 2 Diabetes
Keywords: self monitoring of blood glucose; lancing device; type 2 diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: Each group use lancet (or laser) for first 2 months, take wash out period for 1month, then use laser (or lancet) for another 2 months.
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- laser lancing device (LMT-1000) first user (Experimental): Subjects measure blood glucose using laser lancing device (LMT-1000) for first 2 months, then take a month for wash out period, after that do using lancet for following 2 months.
  Interventions: Device: laser lancing device or lancet for blood glucose level measurement
- lancet first user (Active Comparator): Subjects measure blood glucose using lancet for first 2 months, , then take a month for wash out period, after that do using laser lancing device (LMT-1000) for following 2 months.
  Interventions: Device: laser lancing device or lancet for blood glucose level measurement

INTERVENTIONS:
Device: laser lancing device or lancet for blood glucose level measurement — Subjects measure blood glucose level using laser lancing device (LMT-1000) and lancet for 2 months each.

SUMMARY:
Self monitoring of blood glucose level is crucial in diabetes management, but currently available methods, lancet, have shown low compliance of self monitoring of blood glucose because of pain, keratinization of finger tip, secondary infection. The purpose of this study is evaluating laser lancing device which cause much less pain than lancet to increase compliance of blood sugar checking, and to establish self monitoring system for patients of chronic diseases.

The investigators recruit total of 80 type 2 diabetes patients who visit Korea University Medical center Guro and Ansan hospital. HbA1c level of subject is more than 6.5% and less than 8.5%, and their age is above 20 years and under 80 years. Subjects are randomly distributed in group A or B. Group A subjects use laser device to check blood glucose for 2 months, then take a month for wash out period. After wash out period, participants use lancet for following 2 months. Group B perform the process vice versa. The investigators evaluate the number of blood glucose measurement, HbA1c, diabetes distress scale, average pain score, average satisfaction score from each group.

DETAILED DESCRIPTION:
Self monitoring of blood glucose level is crucial in diabetes management, so it is important to increase compliance of blood glucose checking. Lancet which is currently available methods have shown low compliance of self monitoring of blood glucose, since it causes pain, keratinization of finger tip, secondary infection. The purpose of this study is evaluating laser lancing device which cause much less pain than lancet to increase compliance of blood sugar checking, and to establish self monitoring system for patients of chronic diseases.

The investigators recruit total of 80 subjects who visit Korea University Medical center Guro and Ansan hospital. Study subject are type 2 diabetes whose glycated hemoglobin level is more than 6.5% and less than 8.5%, and whose age is more than 20 years and under 80 years. Subjects are randomly distributed in group A or B. Group A subjects use laser device to check blood glucose for 2 months, then take a month for wash out period. After wash out period, participants use lancet for following 2 months. Group B subjects use lancet first, then have a month for wash out period, after then, switch to laser device afterwards. During washout period, participants use usual glucose checking method which subjects had used. The investigators evaluate the number of blood glucose measurement, glycated hemoglobin, diabetes distress scale, average pain score, average satisfaction score from each group. Also the investigators compare blood glucose, liver function test, lipid level between values from one hand measured by lancet, and values from the other hand measured by laser lancing device.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes patients who visit Korea University medical center, Guro hospital, Ansan hospital
* Patients with Hba1c more than 6.5% and less than 8.5%
* Adults who are able to measure blood glucose level by themselves
* Adults who are able to lance their same finger from both hands
* Adults who comprehend risk of participating in the clinical research, who are able to communicate each other, who are able to follow rules of clinical research
* Subjects who decide to participate in the clinical research voluntarily and sign in the consent format after being informed purposes, methods, expectations of the clinical research

Exclusion Criteria:

* Subject whose age is younger than 19 or older than 80
* students of research institutes
* Pregnant and lactating women
* Subjects who are not able to make decision
* Subjects who are in emergency or being hospitalized
* Subjects who cannot lance sane finger from both hands
* Subjects who are infected by HIV in hospital records
* Subjects who have thrombocytopenia, coagulation disorder or haemophilia
* Subjects who are incompatible for clinical research as researcher evaluated

Ages: 20 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2021-08-10 (Actual); Primary Completion 2022-03-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
average number of checking blood glucose per week | two months after using the device
  Study subject is going to be surveyed about 'average number of checking blood glucose per week' at 2 month after using lancet device, and 2 month after using laser lancing device (LMT-1000)
glycated hemoglobin level | two months after using the device
  Study subject is going to be checked glycated hemoglobin level at 2 month after using lancet device, and 2 month after using laser lancing device (LMT-1000). Data will be shown in percent (%).

SECONDARY OUTCOMES:
average satisfaction score | two months after using the device
  Study subject is going to be surveyed about 'average satisfaction score' at 2 month after using lancet device, and 2 month after using laser lancing device (LMT-1000)
average pain scale | two months after using the device
  Study subject is going to be surveyed about 'average pain scale' at 2 month after using lancet device, and 2 month after using laser lancing device (LMT-1000)
Diabetes Distress Scale | two months after using the device
  Study subject is going to be surveyed about 'Diabetes Distress Scale' at 2 month after using lancet device, and 2 month after using laser lancing device (LMT-1000)
Diabetes Fear of Self-injecting | two months after using the device
  Study subject is going to be surveyed about 'Diabetes Fear of Self injecting' at 2 month after using lancet device, and 2 month after using laser lancing device (LMT-1000)
success rate of measurement of blood glucose by laser lancing device | two months after using the device
  Study subject is going to be surveyed about 'success rate of measurement of blood glucose by laser lancing device' at 2 month after using lancet device, and 2 month after using laser lancing device (LMT-1000)

CONTACTS AND LOCATIONS:
Locations (1):
- Korea University medical center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No